CLINICAL TRIAL: NCT00918333
Title: A Phase I/II Study of the Histone Deacetylase (HDAC) Inhibitor LBH589 (Panobinostat) in Combination With mTOR Inhibitor RAD001 (Everolimus) in Patients With Relapsed Multiple Myeloma or Lymphoma
Brief Title: Panobinostat and Everolimus in Treating Patients With Recurrent Multiple Myeloma, Non-Hodgkin Lymphoma, or Hodgkin Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC0886; NCI-2009-00934 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 08-004746; CLBH589BUS17T; MC0886 (Other: Mayo Clinic); P30CA015083 (NIH); NCT01417559 (obsolete NCT alias)
Record Dates: First submitted 2009-06-01; First posted 2009-06-11 (Estimated); Results first posted 2018-05-18 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; B-cell Adult Acute Lymphoblastic Leukemia; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Hepatosplenic T-cell Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Post-transplant Lymphoproliferative Disorder; Primary Central Nervous System Non-Hodgkin Lymphoma; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Multiple Myeloma; Splenic Marginal Zone Lymphoma; T-cell Adult Acute Lymphoblastic Leukemia; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Hodgkin Disease; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Panobinostat; Everolimus

ARMS (1):
- Treatment (panobinostat and everolimus) (Experimental): Patients receive panobinostat PO QD or on days 1, 3, 5, 15, 17, and 19 and everolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: panobinostat; Drug: everolimus; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: panobinostat — Given PO
  Other Names: Faridak; HDAC inhibitor LBH589; histone deacetylase inhibitor LBH589; LBH589
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of panobinostat and everolimus when given together and to see how well they work in treating patients with multiple myeloma, non-Hodgkin lymphoma, or Hodgkin lymphoma that has come back. Panobinostat and everolimus may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated doses (MTD) of LBH589 (panobinostat) and RAD001 (everolimus) when used in combination in patients with myeloma or lymphoma. (Phase I) II. To evaluate the therapeutic activity of the combination of LBH589 with RAD001 in patients with relapsed or refractory lymphoma. (Arm A, phase II) III. To evaluate the therapeutic activity of the combination of LBH589 with RAD001 in patients with relapsed or refractory multiple myeloma. (Arm B, phase II)

SECONDARY OBJECTIVES:

I. To describe the toxicities associated with the combination of LBH589 with RAD001. (Phase I) II. To further describe the toxicities associated with the combination of LBH589 with RAD001 in each arm independently. (Phase II) III. To evaluate overall survival, progression-free survival, and duration of response in each arm independently. (Phase II)

TERTIARY OBJECTIVES:

I. To evaluate the pharmacokinetic interaction of LBH589 and RAD001. II. To assess the correlation between clinical (toxicity and/or tumor response or activity) effects with the pharmacologic (pharmacokinetic/pharmacodynamic) parameters, and/or biologic (correlative laboratory) results.

OUTLINE: This is a phase I, dose-escalation study of panobinostat and everolimus followed by a phase II study. (dose-escalation closed to accrual as of April 6, 2011)

Patients receive panobinostat orally (PO) once daily (QD) or on days 1, 3, 5, 15, 17, and 19 and everolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Relapsed or refractory multiple myeloma requiring therapy, who have failed, unable to tolerate, or refused other available active therapies
* Biopsy-proven relapsed or refractory non-Hodgkin lymphoma or Hodgkin disease requiring treatment, who have failed, unable to tolerate, or refused other available active therapies; patients should not have other treatment options considered curative; (NOTE: for patients with lymphoma, a re-biopsy is necessary unless the patient has had a previous biopsy < 6 months prior to treatment on this protocol if there has been no intervening treatment; patients with biopsy-proven central nervous system [CNS] lymphoma at any time are not required to have a re-biopsy to be eligible for this study)
* Multiple myeloma:

  * Serum monoclonal protein >= 1.0 g/dL
  * >= 200 mg of monoclonal protein in the urine on 24 hour electrophoresis
  * Serum immunoglobulin free light chain >= 10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
  * Monoclonal bone marrow plasmacytosis >= 30% (evaluable disease) at time of registration
* Lymphoma:

  * Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) or the CT portion of the positron emission tomography (PET)/CT; must have at least one lesion that has a single diameter of >= 2 cm or tumor cells in the blood >= 5 x 10^9/L; skin lesions can be used if the area is >= 2 cm in at least one diameter and photographed with a ruler
* The following disease types are eligible:

  * Transformed lymphomas
  * Diffuse large B cell lymphoma
  * Mantle cell lymphoma
  * Follicular lymphoma grade III
  * Precursor B lymphoblastic leukemia/lymphoma
  * Mediastinal (thymic) large B-cell lymphoma
  * Burkitt lymphoma/leukemia
  * Precursor T-lymphoblastic leukemia/lymphoma
  * Primary cutaneous anaplastic large cell lymphoma
  * Anaplastic large cell lymphoma - primary systemic type
  * Small lymphocytic lymphoma/chronic lymphocytic leukemia
  * Follicular lymphoma, grades 1, 2
  * Extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue (MALT) type
  * Nodal marginal zone B-cell lymphoma
  * Splenic marginal zone B-cell lymphoma
  * Peripheral T cell lymphoma, unspecified.
  * Anaplastic large cell lymphoma (T and null cell type)
  * Lymphoplasmacytic lymphoma (Waldenstrom Macroglobulinemia)
  * CNS lymphoma
  * Post transplant lymphoproliferative disorders
  * Mycosis fungoides/Sezary syndrome
  * Hodgkin Disease
  * Primary effusion lymphoma
  * Blastic natural killer (NK)-cell lymphoma
  * Adult T-cell leukemia/lymphoma
  * Extranodal NK/T-cell lymphoma, nasal type
  * Enteropathy-type T-cell lymphoma
  * Hepatosplenic T-cell lymphoma
  * Subcutaneous panniculitis-like T-cell lymphoma
  * Angioimmunoblastic T-cell lymphoma
  * Anaplastic large cell lymphoma - primary cutaneous type
* For lymphoplasmacytic lymphoma patients without measurable lymphadenopathy, measurable disease can be defined by both of the following criteria:

  * Bone marrow lymphoplasmacytosis with > 10% lymphoplasmacytic cells or aggregates, sheets, lymphocytes, plasma cells, or lymphoplasmacytic cells on bone marrow biopsy and
  * Quantitative immunoglobulin (Ig)M monoclonal protein > 1,000 mg/dL
* Absolute neutrophil count (ANC) >= 1000/uL
* Hemoglobin (Hgb) >= 9 g/dl
* Platelets (PLT) >= 75,000/uL
* Total bilirubin =< 1.5 x upper limit of normal (ULN) or if total bilirubin is > 1.5 x ULN the direct bilirubin must be normal
* Aspartate aminotransferase (AST) =< 3 x ULN
* Creatinine =< 2.5 x ULN
* Serum potassium, magnesium and phosphorus >= lower limit of normal (LLN) and =< 1.2 x ULN
* Ionized calcium >= LLN
* Thyroid-stimulating hormone (TSH) =< 1.5 x ULN; patients are permitted to receive thyroid hormone supplements to treat underlying hypothyroidism
* Ability to understand and the willingness to sign a written informed consent document
* Willingness to return to Mayo Clinic or National Cancer Institute, National Institutes of Health (NIH) - Medical Oncology Branch, Center for Cancer Research (CCR)
* Life expectancy >= 12 weeks
* Willing to provide blood samples for research studies as required by the protocol
* Negative pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2

Exclusion Criteria:

* Candidate for known standard therapy for the patient's disease that is potentially curative
* Uncontrolled infection
* Therapy with myelosuppressive chemotherapy or biologic therapy < 3 weeks unless the patient has recovered from the nadir of the previous treatment to a level that meets the inclusion eligibility criteria of this protocol; NOTE: patients who have received prior RAD001 therapy will be allowed but must meet above requirements
* Receiving corticosteroids > 20 mg of prednisone per day (or equivalent); NOTE: patients may be receiving stable (not increased within the last month) chronic doses of corticosteroids with a maximum dose of 20 mg of prednisone per day if they are being given for disorders other than lymphoma (with the exception of CNS lymphoma, which steroids are permitted at the lowest possible dose necessary and should not be escalated during treatment) such as rheumatoid arthritis, polymyalgia rheumatica or adrenal insufficiency, or asthma
* Persistent toxicities >= grade 2 from prior chemotherapy or biological therapy regardless of interval since last treatment
* Impaired cardiac function or clinically significant cardiac diseases, including any one of the following:

  * Patients with congenital long QT syndrome
  * History or presence of sustained ventricular tachyarrhythmia; (patients with a history of atrial arrhythmia are eligible but should be discussed with the Sponsor prior to enrollment)
  * Any history of ventricular fibrillation or torsade de pointes
  * Bradycardia defined as heart rate (HR) < 50 beats per minute (bpm;) patients with pacemakers are eligible if HR >= 50 bpm
  * Screening electrocardiogram (ECG) with a QTcFredericia (QTcF) > 450 msec
  * Right bundle branch block + left anterior hemiblock (bifascicular block)
  * Patients with myocardial infarction or unstable angina =< 6 months prior to starting study drug
  * Other clinically significant heart disease (e.g., congestive heart failure [CHF] New York [NY] Heart Association class III or IV, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen)
* Any of the following:

  * Pregnant women or women of reproductive ability who are unwilling to use effective contraception
  * Nursing women
  * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational (utilized for a non-Food and Drug Administration [FDA]-approved indication and in the context of a research investigation); NOTE: patients may undergo palliative concurrent radiation of myeloma lesions for pain control or impending fracture, provided the lesion(s) by themselves do not constitute progression
* Known positivity for human immunodeficiency virus (HIV) or hepatitis C with uncontrolled disease; baseline testing for HIV is not required; Note: a detailed assessment of Hepatitis B/C medical history and risk factors must be done at screening for all patients; hepatitis b virus (HBV) deoxyribonucleic acid (DNA) and hepatitis C virus (HCV) ribonucleic acid (RNA) polymerase chain reaction (PCR) testing are required at screening for all patients with a positive medical history based on risk factors and/or confirmation of prior HBV infection
* Active other malignancy requiring treatment that would interfere with the assessments of response of the lymphoma or myeloma to protocol treatment
* Inability to swallow or impairment of gastrointestinal function or gastrointestinal disease that may significantly alter the absorption of the drugs (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection) that would preclude use of oral medications
* Thrombotic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months
* Any severe and/or uncontrolled medical conditions or other conditions that, in the treating physician's opinion, could adversely impact their ability to participate in the study; NOTE: patients on chronic oxygen therapy, those with liver disease such as cirrhosis, chronic hepatitis or chronic persistent hepatitis, or uncontrolled infections will be excluded
* Known hypersensitivity to RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus)
* Receiving any medications or substances that are strong or moderate inhibitors of CYP3A4; receiving any medications or substances that are inducers of CYP3A4
* Using medications that have a relative risk of prolonging the QT interval or inducing torsade de pointes if treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Active bleeding tendency; NOTE: patients on therapeutic anticoagulation should be monitored carefully to maintain therapeutic level of anticoagulation to avoid increased risk of bleeding due to concurrent drug induced thrombocytopenia; it is suggested that patients who require anticoagulation therapy while on therapy use low molecular weight heparin (LMWH)
* Major surgery =< 4 weeks prior to registration or have not recovered from side effects of such therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-06 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mark O Hatfield-Warren Grant Magnuson Clinical Center, Bethesda, Maryland
  - Mayo Clinic, Rochester, Minnesota

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I (Panobinostat + Everolimus): Patients receive 10, 15, 20, 30 or 40 mg/day panobinostat PO 3 times/week or on days 1, 3, 5, 15, 17, and 19 and 5 or 10 mg/day everolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase II (Panobinostat + Everolimus): Patients receive 20,30, or 40 mg/day panobinostat PO on days 1, 3, 5, 15, 17, and 19 and 5 mg/day everolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I (Panobinostat + Everolimus) | Phase II (Panobinostat + Everolimus)
Started | 26 | 98
Completed | 23 | 93
Not Completed | 3 | 5
Not completed — Drug not taken per protocol | 1 | 0
Not completed — Inadequate amount of drugs provided | 1 | 4
Not completed — Ineligible | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I (Panobinostat + Everolimus) | Phase II (Panobinostat + Everolimus) | Total
Number analyzed (Participants) | 23 | 93 | 116
Age, Continuous [Median (Full Range); unit: years] | 61.0 [24.0 to 73.0] | 59.0 [20.0 to 84.0] | 59.5 [20.0 to 84.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 28 | 34
  Male | 17 | 65 | 82
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23 | 93 | 116

OUTCOME MEASURES:

1. Primary Outcome: Number of Phase I Participants With Dose-Limiting Toxicity Events (Phase I)
Description: The Maximum Tolerated Dose (MTD) is defined as the dose level below the lowest dose that induces dose-limiting toxicity (DLT) in at least one-third of patients graded according to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. Dose-limiting toxicities include non-hematologic events graded 3 or higher and deemed at least possibly related to treatment. A total of 6 patients treated at the MTD will be sufficient to identify common toxicities at the MTD. The number of patients reporting a dose-limiting event are reported.
Time Frame: 4 weeks
Population: The overall number of participants analyzed noted above were enrolled in and completed Phase I of the study to determine the maximum tolerated dose (MTD).
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I (Panobinostat + Everolimus)
Number analyzed (Participants) | 23
Participants | 0
Statistical Analysis 1: Comparison: Phase I (Panobinostat + Everolimus); Test type: Superiority or Other; Maximum Tolerated Dose (mg) = 40

2. Primary Outcome: Overall Response Rate (Phase II)
Description: For myeloma, a complete response(CR, defined as Negative immunofixation(IFE) of the serum and urine, < 5% plasma cells in bone marrow(BM), Disappearance of plasmacytomas), stringent CR(sCR, defined as CR plus Normal serum FLC ratio, Absence of clonal cells in BM), very good partial response(VGPR, defined as PR plus Serum and urine M-component detectable by IFE but not on electrophoresis), partial response(PR, defined as a ≥ 50% reduction of serum M-protein and/or reduction in 24-h urinary M-protein by ≥ 90% or to <200 mg per 24 h), or minor response(MR, defined as ≥25% but < 49% reduction of serum M-protein and reduction in 24h urine M-protein by 50-89%) noted as the objective status. For lymphoma, a CR(defined as no evidence of measurable disease), or PR(defined as regression of measurable disease and no new sites of disease) noted as the objective status. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients.
Time Frame: Up to 12 courses
Population: Patients who were enrolled in and completed Phase II and treated at a starting dose of 20 mg or 30/40 mg LBH589 were evaluated in this analysis.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Phase II (Lymphoma Patients Receiving 20 mg LBL589): Lymphoma patients receive 20 mg/day panobinostat (LBH589) PO on days 1, 3, 5, 15, 17, and 19 and 5 mg/day everolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase II (Myeloma Patients Receiving 20 mg LBH589): Myeloma patients receive 20 mg/day panobinostat (LBH589) PO on days 1, 3, 5, 15, 17, and 19 and 5 mg/day everolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase II (Lymphoma Patients Receiving 30/40 mg LBH589): Lymphoma patients receive 30 or 40 mg/day panobinostat (LBH589) PO on days 1, 3, 5, 15, 17, and 19 and 5 mg/day everolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Phase II (Myeloma Patients Receiving 30/40 mg LBH589): Myeloma patients receive 30 or 40 mg/day panobinostat (LBH589) PO on days 1, 3, 5, 15, 17, and 19 and 5 mg/day everolimus PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase II (Lymphoma Patients Receiving 20 mg LBL589) | Phase II (Myeloma Patients Receiving 20 mg LBH589) | Phase II (Lymphoma Patients Receiving 30/40 mg LBH589) | Phase II (Myeloma Patients Receiving 30/40 mg LBH589)
Number analyzed (Participants) | 41 | 14 | 20 | 18
percentage of patients | 39 [23 to 53] | 7 [0 to 34] | 20 [2 to 31] | 0 [0 to 19]

3. Secondary Outcome: Overall Survival Time (Phase II)
Description: Overall survival time is defined as the time from registration to death due to any cause. The median and 95% confidence intervals will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to death due to any cause, assessed up to 2 years post-treatment
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II (Lymphoma Patients Receiving 20 mg LBL589) | Phase II (Myeloma Patients Receiving 20 mg LBH589) | Phase II (Lymphoma Patients Receiving 30/40 mg LBH589) | Phase II (Myeloma Patients Receiving 30/40 mg LBH589)
Number analyzed (Participants) | 41 | 14 | 20 | 18
months | 17.1 [7.0 to NA] — The upper bound of the 95% confidence interval has not yet been reached. | 16.6 [9.7 to NA] — The upper bound of the 95% confidence interval has not yet been reached. | 35.4 [11.5 to NA] — The upper bound of the 95% confidence interval has not yet been reached. | 21.7 [12.1 to 47.6]

4. Secondary Outcome: Progression-free Survival (Phase II)
Description: Progression-free survival time is defined as the time from registration to progression or death due to any cause. Progression is defined for myeloma as Any one or more of the following: Increase of 25% from lowest value in, Serum M-component (absolute increase must be ≥ 0.5 g/dl), Serum M-component increase ≥ 1 g/dl, if lowest M component was ≥ 5 g/dl,Urine M-component (absolute increase must be ≥ 200 mg/24 h), Bone marrow plasma cell percentage (absolute % must be ≥10%) Or any one or more of the following felt related to the underlying clonal plasma cell proliferative disorder: Development of new soft tissue plasmacytomas or bone lesions, Hypercalcemia (≥11.5 mg/dl) Decrease in hemoglobin of ≥2 g/dl, Serum creatinine level ≥2 mg/dl. Progression is defined for lymphoma as any new lesion or increase by ≥50% of previously involved sites from nadir. The median and 95% confidence intervals are estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to progression or death due to any cause, assessed up to 2 years post-treatment
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II (Lymphoma Patients Receiving 20 mg LBL589) | Phase II (Myeloma Patients Receiving 20 mg LBH589) | Phase II (Lymphoma Patients Receiving 30/40 mg LBH589) | Phase II (Myeloma Patients Receiving 30/40 mg LBH589)
Number analyzed (Participants) | 41 | 14 | 20 | 18
months | 3.7 [2.1 to 8.3] | 2.3 [1.0 to NA] — The upper bound of the 95% confidence interval has not yet been reached. | 4.2 [3.0 to 9.6] | 4.3 [3.9 to 5.8]

5. Secondary Outcome: Duration of Response (Phase II)
Description: Duration of response is defined as the time from the date at which the objective status is first noted to be (for myeloma) a complete response (CR, defined as Negative immunofixation(IFE) of the serum and urine, < 5% plasma cells in bone marrow(BM), Disappearance of plasmacytomas), stringent CR(sCR, defined as CR plus Normal serum FLC ratio, Absence of clonal cells in BM), very good partial response(VGPR, defined as PR plus Serum and urine M-component detectable by IFE but not on electrophoresis), partial response(PR, defined as a ≥ 50% reduction of serum M-protein and/or reduction in 24-h urinary M-protein by ≥ 90% or to <200 mg per 24 h) or minor response(MR, defined as ≥25% but < 49% reduction of serum M-protein and reduction in 24h urine M-protein by 50-89%); (for lymphoma) a CR(defined as no evidence of measurable disease), or PR(defined as regression of measurable disease and no new sites of disease) noted as the objective status. Estimated using the method of Kaplan-Meier.
Time Frame: The time from the date at which the patient's objective status is first noted to be a CR, sCR, VGPR, PR, or minor response to the earliest date progression is documented, assessed up to 2 years post-treatment
Population: Patients who were enrolled in and completed Phase II and objective status are first noted to be CR, sCR, VGPR, PR or MR were evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase II (Lymphoma Patients Receiving 20 mg LBL589) | Phase II (Myeloma Patients Receiving 20 mg LBH589) | Phase II (Lymphoma Patients Receiving 30/40 mg LBH589)
Number analyzed (Participants) | 16 | 1 | 4
months | 9.1 [6.5 to 33.5] | NA [NA to NA] — The median and upper bound of the 95% confidence interval have not yet been reached. | 12.9 [4.2 to 30.4]

6. Other Pre Specified Outcome: Change in Pharmacologic (Pharmacokinetic/Pharmacodynamic) Parameters
Description: Changes in parameters will be both graphically and quantitatively summarized and explored. Standard paired comparisons methodologies (paired t-tests, Wilcoxon signed rank tests and Fisher's exact tests for interval, ordinal and nominal level data, respectively) will be used to assess changes in these variables before and after therapy. In addition, these changes in pharmacologic markers and biological results will be explored in relation to clinical outcome to explore any differences between responders and non-responders.
Time Frame: Day 5 and 19 of the first course and then day 1 of each subsequent courses (courses 2-4) prior to the daily dose and 1 and 2 hours after each dose
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Changes in Biological Markers
Description: as for outcome 6
Time Frame: Baseline to up to 12 courses
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed during treatment phase on day 1 of cycles 2-13 and then every 3 cycles; up to 52 months.
Description: CTCAE term (AE description) and grade: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 will be utilized for AE reporting. Each CTCAE term in the current version is a unique representation of a specific event used for medical documentation and scientific analysis and is a single MedDRA Lowest Level Term (LLT).
Arm/Group | Phase I (Panobinostat + Everolimus) | Phase II (Panobinostat + Everolimus)
All-Cause Mortality (participants affected / at risk) | 0/23 | 1/93
Serious Adverse Events (participants affected / at risk) | 3/23 | 25/93
Other Adverse Events (participants affected / at risk) | 23/23 | 92/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (Panobinostat + Everolimus) (N=23) | Phase II (Panobinostat + Everolimus) (N=93)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 0 (0) | 2 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 3 (4)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 5 (6)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum calcium increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Serum triglycerides increased (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash desquamating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I (Panobinostat + Everolimus) (N=23) | Phase II (Panobinostat + Everolimus) (N=93)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 22 (167) | 91 (349)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Keratitis (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 15 (76) | 54 (204)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 16 (71) | 52 (101)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 10 (28) | 41 (112)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (5) | 30 (47)
Chills (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 3 (4)
Fatigue (General disorders) | 21 (126) | 83 (346)
Fever (General disorders) | 0 (0) | 3 (3)
Localized edema (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (3)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (2)
Bone infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 2 (2)
Lip infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Opportunistic infection (Infections and infestations) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 1 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 4 (6) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 2 (4) | 2 (4)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 3 (4)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 2 (2)
Alkaline phosphatase increased (Investigations) | 0 (0) | 6 (10)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 4 (4)
Creatine phosphokinase increased (Investigations) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 0 (0) | 8 (9)
INR increased (Investigations) | 0 (0) | 1 (1)
Leukocyte count decreased (Investigations) | 20 (86) | 69 (156)
Lymphocyte count decreased (Investigations) | 10 (16) | 27 (63)
Neutrophil count decreased (Investigations) | 19 (85) | 66 (159)
Platelet count decreased (Investigations) | 22 (117) | 84 (307)
Serum cholesterol increased (Investigations) | 1 (1) | 3 (5)
Weight loss (Investigations) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 6 (8)
Blood glucose increased (Metabolism and nutrition disorders) | 4 (9) | 7 (10)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Serum albumin decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Serum calcium decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 3 (6) | 21 (40)
Serum potassium decreased (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Serum triglycerides increased (Metabolism and nutrition disorders) | 6 (17) | 8 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (5) | 1 (4)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (9) | 0 (0)
Taste alteration (Nervous system disorders) | 5 (12) | 4 (14)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (4)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 4 (6)
Respiratory tract hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 8 (26) | 28 (49)
Hypotension (Vascular disorders) | 0 (0) | 3 (3)
Thrombosis (Vascular disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes